CLINICAL TRIAL: NCT00546624
Title: GEM 1.5 mg b.i.d. to 4.5 mg b.i.d. Versus Lorazepam in GAD (0777-026)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0777-026; 2007_632
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders | interventions — 7-(1,1-dimethylethyl)-6-(2-ethyl-2H-1,2,4-triazol-3-ylmethoxy)-3-(2-fluorophenyl)-1,2,4-triazolo(4,3-b)pyridazine

INTERVENTIONS:
Drug: MK0777

SUMMARY:
This study will determine the effectiveness of MK0777 GEM versus Lorazepam in the treatment of patients with generalized anxiety disorder.

This is an early phase trial and some specific protocol information is in progress and not publicly available at this time. (Full information is available to trial participants).

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with Generalized Anxiety Disorder
* Women of childbearing potential must use a double-barrier methods of contraception and must have a negative blood pregnancy test at the beginning of the study

Exclusion Criteria:

* History of drug or alcohol abuse
* Have previously participated in another study using MK0777

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2002-11; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC